CLINICAL TRIAL: NCT02434848
Title: A Pilot Study Comparing the Immunogenicity of Fendrix vs. Double-dose Engerix B in HIV-infected Non-responders to Standard Hepatitis B Vaccination Courses
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STH17302
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: HIV; Communicable Diseases; Hepatitis B; HBV; Infectious Diseases
MeSH Terms: conditions — Communicable Diseases; Hepatitis B | interventions — Engerix-B; Fendrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Engerix B (Active Comparator): 15 subjects per group (n = 30 in total)
  Interventions: Drug: Engerix B
- Fendrix (Active Comparator): 15 subjects per group (n = 30 in total)
  Interventions: Drug: Fendrix

INTERVENTIONS:
Drug: Engerix B — Engerix B 20 micrograms/1ml Licensee: GlaxoSmithKline UK Intra-muscular
  Prescription and administration:
  The vaccine will be stored in the Investigators pharmacy as clinical trial stock and dispensed on a subject by subject basis.
  Shelf life and storage The product must be kept refrigerated (2°C - 8°C). Prescriptions will be written and dispensed from pharmacy on the day of consent, screening and vaccination. The shelf life is 3 years.
  Arms: Engerix B
Drug: Fendrix — Fendrix suspension for injection GlaxoSmithKline UK
  Route of Administration, dose regimen:
  Intra-muscular Dose: 0.5ml (20mcg of Hepatitis B Surface Antigen) per vaccination at baseline and weeks 4, 8 and 24.
  Prescription and administration:
  The vaccine will be stored in the Investigators pharmacy as clinical trial stock and dispensed on a subject by subject basis.
  Packaging and labeling The vaccine will have clinical trial labeling. Shelf-life and storage The product must be kept refrigerated (2°C - 8°C).
  The shelf life is 3 years.
  Arms: Fendrix

SUMMARY:
Hepatitis B virus (HBV) infection can result in a greater risk of adverse outcomes in HIV-infected individuals, including more rapid progression to cirrhosis and associated complications such as hepatocellular carcinoma. For this reason, as well as the shared routes of transmission between the two viruses, UK and International guidance recommends that all HBV-negative HIV-infected individuals be offered vaccination against HBV. Unfortunately, response rates in this population can be as low as 17.5 - 40% to standard vaccination courses. To improve this response, strategies such as the use of double dose of standard vaccines (e.g. Engerix B) is recommended in several guidelines for previous non-responders, although there is currently limited evidence for this approach. An alternative strategy is to use vaccines with novel adjuvants such as Fendrix and observational clinical data in the Investigators HIV cohort suggests that response rates can be as high as 81% of individuals achieving HBV surface antibody (HBsAb) levels >100 in a group that did not respond to previous standard HBV vaccine courses. However, the cost of Fendrix is considerably higher than Engerix B and controlled trials are required to confirm whether this approach is warranted. Furthermore, insights into the potential mechanisms by which Fendrix may elicit better responses would be valuable in optimising future vaccine strategies in this population.

The Investigators propose to conduct a randomised, open label, active-controlled pilot study comparing double dose Engerix B and Fendrix in HIV-infected non-responders to standard HBV vaccine courses, which will provide the necessary data to design and power a larger multicentre randomised controlled trial. Outcome measures will include the proportion of individuals seroconverting with HBsAb levels >100 following each vaccination course, the magnitude and quality of the HBV-specific CD4+ T-cell responses elicited by each vaccine and the durability of the HBsAb response at 1 year following the end of vaccination.

DETAILED DESCRIPTION:
To compare the immunological responses in HIV-infected non-responders to standard hepatitis B vaccination courses to immunization with either double-dose Engerix B or Fendrix:

1. Investigators will measure the proportion of individuals seroconverting with Hepatitis B surface antibody titres of >100 (and ≥10) IU/ml at 8 weeks after the immunisation course, as well as the durability of this response at 1 year following the completion of the course. The primary aim will be to provide some preliminary data from a head to head study of these two approaches with which to power a larger multi-centre randomized controlled trial.
2. Investigators will define the magnitude and quality of the Hepatitis B-specific CD4+ T-cell response following vaccination, thus obtaining key immunological data to fill the knowledge gap in T-cell responses to Hepatitis B vaccination, required to support the rationale design of future multi-centre, randomized study comparing vaccination strategies in HIV-infected non-responders to standard Hepatitis B vaccine courses.

The research is original. There is only one published study to date looking at the efficacy of double-dose Engerix B in HIV-infected non-responders to standard courses1. There is currently anecdotal experience of the use of Fendrix in this group from the Investigators cohort and others. There are no head-to-head comparisons of these two strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* HIV-1 infected
* On antiretroviral therapy
* Viral load undetectable (for at least 6 months, last available measurement within 3 months)
* History of having received at least one complete course of non-Fendrix-based hepatitis B vaccination in the past. Patients who have already received a double-dose Engerix B course in the past will still be eligible.
* HBsAb levels persistently <10IU/L despite vaccination

Exclusion Criteria:

* A history of hypersensitivity to any previous hepatitis B vaccination
* A history of hypersensitivity to any components of either Engerix B or Fendrix (see Summary of Product Characteristics).
* Currently undergoing an incomplete course of any hepatitis B vaccination
* Having received at least one vaccination with Fendrix in the past
* Recipient of any other vaccination within the last 2 weeks
* Any previously detectable HBsAb level (≥10)
* Pregnant or breastfeeding
* Individuals who have a current severe febrile illness
* Individuals with a known and current history of anaemia or any symptoms (shortness of breath, chronic fatigue, chest pain or pallor) suggestive of possible anaemia or haemoglobin below the lower limit of sex adjusted normal range on a full blood count taken within the last 3 months.
* Current (active) participation in any clinical trial
* Inability to communicate in English or convey willingness to participate
* End Stage Renal Disease undergoing renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
The proportion of individuals seroconverting with Hepatitis B surface antibody titres of >100 (and ≥10) IU/ml | 8 weeks

SECONDARY OUTCOMES:
Hepatitis B-specific CD4+ T-cell response at 2 weeks following the first vaccination and 2 weeks following the 3rd vaccination. | 2 weeks following the first vaccination and 2 weeks following the 3rd vaccination.
The proportion of individuals seroconverting with Hepatitis B surface antibody titres of >100 (and ≥10) IU/ml | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom